CLINICAL TRIAL: NCT02991963
Title: Epidemiology of Malaria in Ubon Ratchathani, Thailand: a Case-control Study
Brief Title: Epidemiology of Malaria in Ubon Ratchathani, Thailand
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Oxford (Other)
Collaborators: Mahidol Oxford Tropical Medicine Research Unit (Other)
Responsible Party: Sponsor
Other Study IDs: EPI1601
Record Dates: First submitted 2016-12-09; First posted 2016-12-14 (Estimated); Last update posted 2017-01-20 (Estimated); Status verified 2017-01

CONDITIONS: Epidemiology
MeSH Terms: interventions — Interviews as Topic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — 1. Dried Blood Spot
     * To extract information on a broad variety of genetic variations.
     * To analyse for P. falciparum multi-drug resistance gene (MDR) copy number as a marker of mefloquine resistance, as well as for merozoite surface protein (MSP), glutamate rich protein (GLURP) and other markers to compare with follow-up samples to identify relapses and recrudescences.
  2. Venous Blood for parasite culture and in vitro drug sensitivity, cryopreservation of parasites, malaria immunological tests, antimalarial pharmacokinetics, ultrasensitive Plasmodium PCR and whole genome sequencing
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Case: Malaria patient defined by positive RDT or blood smear
  Interventions: Other: Interview; Other: Blood collection (Dried Blood Spot); Other: Blood Collection (Venous Blood collection); Other: Blood Smear
- Control: Non-malaria patient defined by negative RDT or blood smear
  Interventions: Other: Interview; Other: Blood Collection (Venous Blood collection); Other: Blood Smear

INTERVENTIONS:
Other: Interview — A survey will be included patient demographics, information on malaria treatment, bed net use and possible risk factors for acquiring malaria, as well as questions about their travel and usage of mobile phones
Other: Blood collection (Dried Blood Spot) — Dried Blood Spot
  Groups: Case
Other: Blood Collection (Venous Blood collection) — Venous Blood collection
Other: Blood Smear — Slide blood smear

SUMMARY:
This is an observational study (case-control study) aiming to identify risk factors for malaria infection in health centers or malaria posts or district hospitals in Buntharik District and Nachalui District, Ubon Ratchathani Province, Thailand.

This study expects to recruit 330 cases (malaria positive) and 330 control (negative cases) subject. One-to-one matching of cases (malaria positive) and controls (malaria negative) will be done at each study site.

CASE (Malaria positive) subject will go through the following;

1. Enrollment visit (Day 0)

   1.1 Blood collection of three dried blood spots, and malaria slide. In district hospitals in individuals >14 kg: additional 10ml venous blood will be collected.

   1.2 A survey questionnaire which includes patient demographics, information on malaria treatment, bed net use and possible risk factors for acquiring malaria, as well as questions about their travel and usage of mobile phones will be administered.
2. Follow up visits (if fever plus Day 42 (+/-3))

2.1 Blood collection of three dried blood spots and malaria slide. In district hospitals: additional 0.5ml venous blood will be collected.

2.2 Short survey questionnaire including questions on symptoms, travel and possible risk behaviors since enrollment will be administered.

CONTROL (Malaria negative) subject will go through the following;

1. Enrollment visit (Day 0)

   1.1 Blood collection to confirm negative malaria slide. In district hospitals: additional 0.5ml venous blood will be collected.

   1.2 A survey questionnaire including patient demographics, information on any recent malaria treatment they may have taken, bed net use and possible risk factors for acquiring malaria, as well as questions about their travel and usage of mobile phones will be administered.
2. Follow up visit: No follow up visit

DETAILED DESCRIPTION:
Study sites and enrollment:

Patients self-presenting to (1) health centres or(2) malaria posts or (3) district hospitals in Buntharik District and Nachalui District, Ubon Ratchathani Province, Thailand and requiring a diagnostic test for malaria as determined by the treating clinician will be recruited. Those who are malaria positive will be candidate cases and those who are malaria negative will be candidate controls.

One-to-one matching of cases and controls will be done at each study site. One control will be matched to each case. The matching criteria will be the next malaria negative patient to attend the study site of the same gender and age+/-5 years as an enrolled malaria positive case.

Study procedure:

CASE (Malaria patient defined by positive RDT or blood smear)

Upon enrollment, the below study procedures will be followed;

1. Blood samples consisting of:

   * Three dried blood spots
   * A microscopy slide
   * In the district hospitals only, 10 ml of venous blood will be taken from the positive for malaria patient.
2. A survey include patient demographics, information on malaria treatment, bed net use and possible risk factors for acquiring malaria, as well as questions about their travel and usage of mobile phone will be administered to each patient.

CONTROL (Non-malaria patient defined by negative RDT or blood smear)

Upon enrollment, for those negative for malaria, the below study procedures will be follows;

1. Blood samples consisting of:

   * Blood smear
   * In the district hospitals only, 0.5 ml of venous blood will also be collected.
2. A survey include patient demographics, information on malaria treatment, bed net use and possible risk factors for acquiring malaria, as well as questions about their travel and usage of mobile phone swill be administered to each patient.

CASE: Follow-up

* If patients develop a fever after the end of antimalarial treatment and within 42 days after enrollment, they will be asked to return for follow-up as soon as possible on one occasion and then again at 42 (+/-3) days.
* If they do not develop fever within 42 days after enrollment, they will be asked to return for follow up at 42 (+/-3) days.

At the follow-up visit, blood will be taken to test for malaria by microscopy, three dried blood spots will be taken and a short survey administered including questions on symptoms, travel and possible risk behaviors since enrollment.

*In the district hospitals only, 1.5ml of venous blood will be taken

CONTROL: No follow up

ELIGIBILITY:
Inclusion Criteria:

- Case (Malaria patient defined by positive RDT or blood smear):

* Patients of ≥ 6 months of age testing positive for malaria of any species as determined by a positive rapid diagnostic test (RDT) or asexual stage parasites on a smear of peripheral blood including individuals with more than one species of Plasmodium.

  * Control (Non-malaria patient defined by negative RDT or blood smear):
* Patients > 6 months of age requiring a diagnostic test for malaria but testing negative for malaria by rapid diagnostic test (RDT) or asexual stage parasites on a smear of peripheral blood. Controls will be age and gender matched to individual cases at each study site (details below).

Exclusion Criteria:

Not willing to provide written informed consent.

Min Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients self-presenting to health centres or malaria posts or district hospitals in Buntharik District and Nachalui District, Ubon Ratchathani Province, Thailand and requiring a diagnostic test for malaria as determined by the treating clinician will be recruited. Those who are malaria positive will be candidate cases and those who are malaria negative will be candidate controls.
Sampling Method: Non-Probability Sample
Enrollment: 660 (Estimated)
Dates: Start 2016-12 (Actual); Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Risk factors for Malaria infection | 2 years
  Risk factors for malaria infection in Ubon Ratchathani Province, Thailand

SECONDARY OUTCOMES:
Proportion of malaria infections in Ubon Ratchathani Province | 2 years
  Proportion of malaria infections that are imported in Ubon Ratchathani Province, Thailand
Prevalence of clinical antimalarial drug resistance | 2 years
  Prevalence of clinical antimalarial drug resistance in cases of P. falciparum malaria in Ubon Ratchathani Province, Thailand
Human movement leading to spread of malaria and antimalarial drug resistance | 2 years
  4. Estimates of the potential for spread of malaria and antimalarial drug resistance from Ubon Ratchathani Province, Thailand through human movement to other locations.
Measure antimalarial drug in blood prior to participate in the study | 2 years
  List of antimalarials which patients have recently taken, if any, prior to presentation in order to estimate drug pressure on the parasite population.

CONTACTS AND LOCATIONS:
Locations (1):
- Buntharik Hospital, Ubon Ratchathani, Ubon Rachatani, Thailand

IPD SHARING:
Plan to Share IPD: Yes
According to Mahidol-Oxford Tropical Medicine Research Unit policy